CLINICAL TRIAL: NCT05540730
Title: Analysis of Foot Plantar Pressure Behavior of Children With Obstetric Brachial Plexus Paralysis
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Yunus Özdemir, PhD, Dr, Istanbul Medipol University Hospital
Other Study IDs: IstanbulMUH-DPTR-Yozdemir-0094
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Brachial Plexus Palsy; Gait Disorders in Children
Keywords: Brachial Plexus Palsy; Gait Disorders in Children; Biomechanics; Gait Analysis
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstetric brachial plexus paralysis
  Interventions: Diagnostic Test: Gait Analysis
- Control
  Interventions: Diagnostic Test: Gait Analysis

INTERVENTIONS:
Diagnostic Test: Gait Analysis — Foot plantar pressure with pedobarography and arm swing with video camera will be analyzed.

SUMMARY:
The aim of this study was to investigate the foot plantar pressure behavior alterations during gait for children with obstetric brachial plexus (OBBP). 19 children with OBBP and 10 healthy children will be included in the study. The inclusion criteria of the study were to be between the ages of 7-15, not have a history of surgery or botox in the last 6 months, and not have any other disease. Foot plantar pressures of all participants will be analyzed with a pedobarography device. For arm swing analysis, a video camera will be recorded during walking and arm flexion/extension angles will be measured with Kinovea software.

ELIGIBILITY:
Inclusion Criteria:

- Between the ages of 7-15. No other disease

Exclusion Criteria:

- Having undergone surgery or botox intervention for orthopedic problems in the last 6 months.

Having health problems in the unaffected extremity or adversely affecting general body health.

The participant's parent has not signed the consent form.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with obstetric brachial plexus paralysis
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Stance Time | during gait analysis.
  stance time phase during walking

SECONDARY OUTCOMES:
Step Length | during gait analysis.
Ground reaction force | during gait analysis.
Single limb support phase | during gait analysis.
  Single limb support phase during walking

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No